CLINICAL TRIAL: NCT06926517
Title: Life and Death Issues in the Post-epidemic Era - Life and Death Care, Reflection and Teaching Practice Integrating New Coronavirus Pneumonia Issues
Brief Title: Life and Death Care, Reflection and Teaching Practice Integrating New Coronavirus Pneumonia Issues
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 202400049B0
Record Dates: First submitted 2025-04-07; First posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2024-10

CONDITIONS: Life and Death
Keywords: Life and Death Issues; Post-Epidemic Era
MeSH Terms: conditions — Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- life and death care (Experimental): Life and death issues in the post-epidemic era - Curriculum planning that integrates life and death care, reflective learning and teaching practice on the new coronavirus pneumonia issue, introducing 18-week theme courses, each course is 100 minutes
  Interventions: Other: life and death courses

INTERVENTIONS:
Other: life and death courses — Life and death issues in the post-epidemic era - Curriculum planning that integrates life and death care, reflective learning and teaching practice on the new coronavirus pneumonia issue, introducing 18-week theme courses, each course is 100 minutes

SUMMARY:
The basics of life and death are further extended and can meet the life and death needs of clinical care, which is a breakthrough in the existing life and death courses and innovation. The research purposes of this article are (1) to develop a teaching plan for the "Life and Death Issues in the Post-Epidemic Era" course that incorporates the issue of COVID-19; (2) to explore the implementation process and qualitative and quantitative learning effects of "Life and Death Issues in the Post-Epidemic Era"; ( 3) Understand the researcher's reflections on teaching practice through learning reflection and learning effectiveness analysis results. The teaching methods used in this course include: teacher lectures, non-verbal and affective activities with expressive art media, learning by doing and "hands-on", audio-visual teaching, case studies and group discussions, collaborative teaching with teachers, and reflection. The researchers tried to use reflective theory and practice in course teaching, and through reflective writing exercises on issues, cultivate nursing students' understanding of life and death issues, face their own life attitude, death attitude and self-care, and acquire the basic ability of life and death care.

DETAILED DESCRIPTION:
The world has been affected by the coronavirus for more than four years, with more than 400 deaths. Thousands of people die from the epidemic, which is an almost inevitable death issue for medical staff. However, nursing students lack internship experience and do not have enough opportunities to contact dying patients. They are faced with the sudden death of patients due to the outbreak and limited medical equipment. sex, the medical ethical choices that arise, and the impact on society and the medical field. In the past, life and death courses did not specifically discuss life and death issues related to the epidemic. Therefore, integrating current affairs issues related to the new crown epidemic can help us discuss the existing life and death issues. The basics of life and death are further extended and can meet the life and death needs of clinical care, which is a breakthrough in the existing life and death courses and innovation. The research purposes of this article are (1) to develop a teaching plan for the "Life and Death Issues in the Post-Epidemic Era" course that incorporates the issue of COVID-19; (2) to explore the implementation process and qualitative and quantitative learning effects of "Life and Death Issues in the Post-Epidemic Era"; ( 3) Understand the researcher's reflections on teaching practice through learning reflection and learning effectiveness analysis results. The teaching methods used in this course include: teacher lectures, non-verbal and affective activities with expressive art media, learning by doing and "hands-on", audio-visual teaching, case studies and group discussions, collaborative teaching with teachers, and reflection. The researchers tried to use reflective theory and practice in course teaching, and through reflective writing exercises on issues, cultivate nursing students' understanding of life and death issues, face their own life attitude, death attitude and self-care, and acquire the basic ability of life and death care.

ELIGIBILITY:
Inclusion Criteria:

* Students who are willing to participate in this study and have taken courses in life and death

Exclusion Criteria:

* none

Ages: 20 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Nursing life and death professional knowledge | Tests for the first and eighteenth weeks of the course
  Based on the evaluation of end-of-life diseases (top ten non-cancer) and COVID-19's well-being indications and end-of-life symptoms Assessment and care, the grief and needs of dying patients and their families, the cultural, social and psychological significance and functions of funeral rituals, 20 knowledge test questions on funeral culture and religious healing behaviors of various religions and medical ethics and moral dilemmas, etc.
life attitude scale | Tests for the first and eighteenth weeks of the course
  This study used the short version of the Life Attitude Scale to measure students' attitude towards life before and after the course (Xie and Pan, 2015). The scale includes six dimensions, namely: ideals, autonomy, love and care, and sense of existence. , death attitude, life experience, each aspect has four questions, for a total of twenty-four questions. Score on a Likert-7 scale, with 1 representing strongly disagree and 7 representing strongly agree. The higher the score, the more positive the subject's life attitude. The reference for the integrity of this scale (Xie and Pan, 2015) is Cronbach's α value of 0.93. The results of confirmatory factor analysis found that the theoretical model of the study has a good fit, χ²(237) = 1078.58, χ²/df = 4.55, GFI = 0.93, CFI = 0.93, RMSEA = 0.053.
death attitude scale | Tests for the first and eighteenth weeks of the course
  This study used the Death Attitude Scale, using the revised Wong, Reker and Gesser Death Attitude Description Scale. which contains The sub-scale includes death fear (7 questions), death avoidance (5 questions), neutral acceptance (5 questions), approach-oriented death acceptance (10 questions), and escape acceptance (5 questions); death fear refers to the fear of death. and negative thoughts and feelings about dying; death avoidance refers to a defense mechanism that keeps death in the personal subconscious; the concept of neutral acceptance is the degree to which an individual believes that death is neither feared nor expected; approach-oriented death acceptance It refers to the extent to which an individual sees death as a means to a happy afterlife; avoidance acceptance refers to the extent to which an individual sees death as an escape from a painful existence. Score it on a Likert-5 scale, with 1 representing strongly disagree and 5 representing strongly agree.
Self-compassion scale | Tests for the first and eighteenth weeks of the course
  This time we use Lai Zhichao and Su Lunhui (2015) translated as the Chinese version of the Self-Compassion Scale, the revised Chinese version of the scale has 25 items, with a five-point Likert scale, where 1 means almost never, 5 means almost always, and the score The higher the value, the more consistent it is with the item. It contains three aspects and six mutually opposing factors, divided into positive self-care ability (three groups) and negative self-care ability (three groups), namely: self-kindness-self-criticism (a total of 10 questions), shared suffering- Isolated experiences (8 questions in total) and mindfulness-over-identification (7 questions). The Cronbach's α coefficient of the reference Chinese version of the scale is 0.91, and the component reliability of its three scales (self-kindness, shared suffering, and mindfulness) ranges from 0.85 to 0.88. Validity model fit index: CFI value is 0.97, TLI value is 0.96, RMSEA value is 0.06, and SRMR value is 0.06 .
Spiritual Care Scale | Tests for the first and eighteenth weeks of the course
  The original scale was compiled by Lay Hwa Tiew (2012). The spiritual care-giving scale has 35 questions and 4 facets. The first facet is "Characteristics of spiritual care" (No. 22, 23 , 24, 25, 26, 27, 28, 29, 30, 31, 32, 34 and 35 questions); the second aspect "Spirituality and Definition of Spirit" (No. 6, 15, 16, 17, 18, 19 , 20 and 21 items); five items related to the third facet "spiritual perspective" (items 1, 2, 3, 4 and 5) and the fourth facet "spirituality and spiritual care values" (items 7 , 8, 9, 10, 11, 12, 13 and 14 items). It is scored using a six-point method (1-6 points). The higher the score, the higher the Cronbach's a of the four aspects of the original scale. are 0.94, 0.85, 0.84 and 0.86 (Hu et al., 2019). Before using this scale, it is planned to recruit 400 nursing students through snowballing and convenience sampling to establish the reliability and validity of the scale and make revisions.
Spiritual Health Scale-short version | Tests for the first and eighteenth weeks of the course
  There are 24 questions and 5 facets. Each facet is "Connecting with People" (Questions 1 to 4).Questions), "Live with meaning" (Questions 5 to 10), "Beyond adversity" (Questions 11 to 16), "Religious sustenance" (Questions 17 to 20), "Understand one's own mind " (Questions 21 to 24). The Cronbach's a value of the full scale is 0.93. After factor analysis, the Cronbach's a value of each scale ranges from 0.75 to 0.92. The test-retest reliability after three weeks is 0.77 (Xiao and Huang, 2005).

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Medical Foundation, Tainan, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ruiz-Fernandez MD, Ramos-Pichardo JD, Ibanez-Masero O, Carmona-Rega MI, Sanchez-Ruiz MJ, Ortega-Galan AM. Professional quality of life, self-compassion, resilience, and empathy in healthcare professionals during COVID-19 crisis in Spain. Res Nurs Health. 2021 Aug;44(4):620-632. doi: 10.1002/nur.22158. Epub 2021 May 25. PMID 34036600
- [Background] Pattison N. End-of-life decisions and care in the midst of a global coronavirus (COVID-19) pandemic. Intensive Crit Care Nurs. 2020 Jun;58:102862. doi: 10.1016/j.iccn.2020.102862. Epub 2020 Apr 2. No abstract available. PMID 32280052
- [Background] Pehlivan S, Lafci D, Vatansever N, Yildiz E. Relationship Between Death Anxiety of Turkish Nurses and Their Attitudes Toward the Dying Patients. Omega (Westport). 2020 Nov;82(1):128-140. doi: 10.1177/0030222819895122. Epub 2019 Dec 19. PMID 31856657
- [Background] Cheng L, Guo X, Liu H, Chen Q, Cui R. Hope, death anxiety and simplified coping style scores of nursing students during the outbreak of COVID-19: A cross-sectional study. Medicine (Baltimore). 2021 Aug 27;100(34):e27016. doi: 10.1097/MD.0000000000027016. PMID 34449474
- [Background] Akat, M., Karataş, K. (2020). Psychological effects of COVID-19 Pandemic on society and its reflections on education. Turkish Studies, 15(4), 1-13.